CLINICAL TRIAL: NCT00873080
Title: Reliability of the Angle Measurement of the Software for Photogrammetry Postural Assessment
Brief Title: Reliability of the Angle Measurement of the Software for Photogrammetry Postural Assessment (SAPO)
Acronym: SAPO
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Juliana Alves Souza, University of Santa Maria
Other Study IDs: UFSantaMaria
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Body Posture Alignment Condition; Temporomandibular Disorder
Keywords: reliability; photogrammetry
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study aims to verify the reliability of intra and inter-examiner of angular measures proposed by SAPO postural assessment software. Methods: 24 subjects were photographed and three experienced examiners analyzed the images.

DETAILED DESCRIPTION:
The body posture in the orthostatic position has been widely utilized as in the clinical practice as in the research, for the diagnosis and physiotherapy treatment planning. The photogrammetry has been used as a valuable resource for the physiotherapist's diagnosis and verification of measuring postural changes, but the lack of standardization of anatomic references, the used angles between them and their meaning embarrasses comparison among studies.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years old
* diagnosis of temporomandibular disorder

Exclusion Criteria:

* neurological diseases
* systemic diseases
* lower limbs fracture
* balance disorder

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 24 subjects with temporomandibular disorder
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J A Souza, Principal Investigator — Universidade Federal de Santa Maria